CLINICAL TRIAL: NCT05116488
Title: Detection of Electrocardiographic Brugada Patterns Using High Precordial Leads Positioning Among Asymptomatic Upper Egyptian Population
Brief Title: Detection of Electrocardiographic Brugada Patterns Using High Precordial Leads
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Rashad Ali, Doctor, Assiut University
Other Study IDs: ECG Brugada patterns
Record Dates: First submitted 2021-10-16; First posted 2021-11-11 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Brugada ECG Patterns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ECG(electrocardigraph) — Detection of electrocardiographic Brugada patterns using high precordial leads positioning as placing the precordial leads in the second intercostal space has been proposed to add sensitivity to the ECG diagnosis of Brugada syndrome.

SUMMARY:
Detection of prevalence of Brugada patterns in our locality in asymptomatic patients , by standard 12 lead ECG level and high precordial ECG level, measuring how much the high precordial leads is more sensitive in Brugada patterns detection than standard level 12 lead ECG in our upper Egyptian population.

DETAILED DESCRIPTION:
Detection of prevalence of Brugada patterns in our locality in asymptomatic patients , by standard 12 lead ECG level and high precordial ECG level, measuring how much the high precordial leads is more sensitive in Brugada patterns detection than standard level 12 lead ECG in our upper Egyptian population.

The study will include patients fulfilling our criteria presenting to cardiology outpatient clinic and emergency room of Assiut University hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. patients with IHD,HTN,DM with no organic heart disease by ECHO.
2. healthy persons with normal structure heart by ECHO.

Exclusion Criteria:

1. Acute coronary syndrome.
2. cardiomyopathy.
3. severe valvular heart disease.
4. HTN heart disease with LVH.
5. Malignancy.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include patients fulfilling our criteria presenting to cardiology outpatient clinic and emergency room of Assiut University hospitals.
  All patients will be subjected to:
  A. Full history taking: including age, sex, history of DM, HTN, Smoking, dyslipidaemia symptoms of heart failure, symptoms of Coronary artery disease, and history of any previous arrhythmia.
  B. Full Physical examination:
  * General examination Systolic and diastolic blood pressure and heart rate assessment.
  * Cardiac examination. C. Laboratory investigations: electrolytes ( to make sure they are within normal).
  D. Standard 12lead ECG. E .High precordial ECG: to increase sensitivity of Brugada patterns detection. F. Echocardiography: to exclude structural heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of electrocardiographic Brugada patterns using high precordial leads positioning among asymptomatic upper Egyptian population | up to 4 hours for each case to make sure of meeting eligibility criteria
  Detection of prevalence of Brugada patterns in our locality in asymptomatic patients , by standard 12 lead ECG level and high precordial ECG level, measuring how much the high precordial leads is more sensitive in Brugada patterns detection than standard level 12 lead ECG in our upper Egyptian population.

SECONDARY OUTCOMES:
Follow up of positive cases | six months after diagnosis of Brugada pattern for each case
  The positive cases will be educated regarding their condition, asked about their history of syncope and family history of sudden cardiac death and will be educated about avoiding and rapid management of fever and electrolyte disturbances and educated about the list of drugs to be avoided.
  The positive cases will be followed up for 6 months both clinically and by Holter at 1st, and 6th month for detection of subclinical ventricular arrhythmias.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Eldin Sayed Atta, Professor, Study Director — Assiut University; Mahmoud Abdelsabour, Lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Wilde AA, Antzelevitch C, Borggrefe M, Brugada J, Brugada R, Brugada P, Corrado D, Hauer RN, Kass RS, Nademanee K, Priori SG, Towbin JA; Study Group on the Molecular Basis of Arrhythmias of the European Society of Cardiology. Proposed diagnostic criteria for the Brugada syndrome: consensus report. Circulation. 2002 Nov 5;106(19):2514-9. doi: 10.1161/01.cir.0000034169.45752.4a. No abstract available. PMID 12417552
- [Background] Peritz DC, Chung EH. Criteria for evaluating rSr' patterns due to high precordial ECG lead placement accurately confirm absence of a Brugada ECG pattern. J Electrocardiol. 2016 Mar-Apr;49(2):182-6. doi: 10.1016/j.jelectrocard.2015.12.015. Epub 2016 Jan 6. PMID 26850497
- [Background] Kapplinger JD, Tester DJ, Alders M, Benito B, Berthet M, Brugada J, Brugada P, Fressart V, Guerchicoff A, Harris-Kerr C, Kamakura S, Kyndt F, Koopmann TT, Miyamoto Y, Pfeiffer R, Pollevick GD, Probst V, Zumhagen S, Vatta M, Towbin JA, Shimizu W, Schulze-Bahr E, Antzelevitch C, Salisbury BA, Guicheney P, Wilde AA, Brugada R, Schott JJ, Ackerman MJ. An international compendium of mutations in the SCN5A-encoded cardiac sodium channel in patients referred for Brugada syndrome genetic testing. Heart Rhythm. 2010 Jan;7(1):33-46. doi: 10.1016/j.hrthm.2009.09.069. Epub 2009 Oct 8. PMID 20129283
- [Background] Antzelevitch C, Brugada P, Borggrefe M, Brugada J, Brugada R, Corrado D, Gussak I, LeMarec H, Nademanee K, Perez Riera AR, Shimizu W, Schulze-Bahr E, Tan H, Wilde A. Brugada syndrome: report of the second consensus conference: endorsed by the Heart Rhythm Society and the European Heart Rhythm Association. Circulation. 2005 Feb 8;111(5):659-70. doi: 10.1161/01.CIR.0000152479.54298.51. Epub 2005 Jan 17. PMID 15655131
- [Background] Patel SS, Anees S, Ferrick KJ. Prevalence of a Brugada pattern electrocardiogram in an urban population in the United States. Pacing Clin Electrophysiol. 2009 Jun;32(6):704-8. doi: 10.1111/j.1540-8159.2009.02354.x. PMID 19545330
- [Background] Bachman JW, Field CS, Hammersley CE. Educational program for premature labor. J Am Board Fam Pract. 1992 Nov-Dec;5(6):645-7. No abstract available. PMID 1462800
- [Background] Chung EH. Brugada ECG patterns in athletes. J Electrocardiol. 2015 Jul-Aug;48(4):539-43. doi: 10.1016/j.jelectrocard.2015.05.001. Epub 2015 May 8. PMID 26026871
- [Background] Sangwatanaroj S, Prechawat S, Sunsaneewitayakul B, Sitthisook S, Tosukhowong P, Tungsanga K. New electrocardiographic leads and the procainamide test for the detection of the Brugada sign in sudden unexplained death syndrome survivors and their relatives. Eur Heart J. 2001 Dec;22(24):2290-6. doi: 10.1053/euhj.2001.2691. PMID 11728150
- [Background] Meregalli PG, Wilde AA, Tan HL. Pathophysiological mechanisms of Brugada syndrome: depolarization disorder, repolarization disorder, or more? Cardiovasc Res. 2005 Aug 15;67(3):367-78. doi: 10.1016/j.cardiores.2005.03.005. PMID 15913579
- [Derived] Ali AR, Abdelsabour M, Atta S. Yield of regular practice of high precordial leads electrocardiogram among asymptomatic upper Egyptian population considering Brugada patterns, a cross-sectional study. Egypt Heart J. 2026 Jan 12;78(1):4. doi: 10.1186/s43044-026-00714-x. PMID 41524999